CLINICAL TRIAL: NCT01955213
Title: Clinical Evaluation of the Efficacy of Methylnaltrexone in Resolving Constipation Induced by Different Opioid Subtypes, Combined With Laboratory Analysis of Immunomodulatory and Antiangiogenic Effects of Methylnaltrexone
Brief Title: Methylnaltrexone for Opioid Induced Constipation
Acronym: RILAX
Status: Terminated | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Stichting Nuts Ohra (Other)
Responsible Party: Principal Investigator, H.M.W. Verheul, Prof. dr., Amsterdam UMC, location VUmc
Other Study IDs: 2012/169; 2012-000850-75 (EudraCT Number)
Record Dates: First submitted 2012-12-11; First posted 2013-10-07 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-07

CONDITIONS: Constipation
Keywords: constipation, methylnaltrexone, opoid
MeSH Terms: conditions — Constipation | interventions — methylnaltrexone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — From patients who also give informed consent for the second part of the study 50 ml of heparinized blood will be drawn before the first administration of methylnaltrexone (day 0), after 24 hours (day 1), at day 14 and approximately day 42 for immuno- and angiogenic measurements (see flow chart below).
  From this blood sample the size, phenotype and function of various leukocyte subsets, serum cytokine levels, VEGF levels, thrombocyte levels and circulating endothelial cell levels will be determined by means of fluorescence-activated cell sorting (FACS) or enzyme-linked immunosorbent assay (ELISA).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Morphine Sulphate: Patient groups are defined by the type of opioid used, being either morphine sulphate, fentanyl or oxycodone.Patients will be treated with methylnaltrexone in a standard dosing regimen for their weight: 38-62kg:8 mg, 62-114kg:12 mg, >114 kg: 0.15 mg/kg) Methylnaltrexone will be administered subcutaneously every other day for up to 7 doses.
  Interventions: Drug: methylnaltrexone
- Fentanyl: Patient groups are defined by the type of opioid used, being either morphine sulphate, fentanyl or oxycodone.Patients will be treated with methylnaltrexone in a standard dosing regimen for their weight: 38-62kg:8 mg, 62-114kg:12 mg, >114 kg: 0.15 mg/kg) Methylnaltrexone will be administered subcutaneously every other day for up to 7 doses.
  Interventions: Drug: methylnaltrexone
- Oxycodone: Patient groups are defined by the type of opioid used, being either morphine sulphate, fentanyl or oxycodone.Patients will be treated with methylnaltrexone in a standard dosing regimen for their weight: 38-62kg:8 mg, 62-114kg:12 mg, >114 kg: 0.15 mg/kg) Methylnaltrexone will be administered subcutaneously every other day for up to 7 doses.
  Interventions: Drug: methylnaltrexone

INTERVENTIONS:
Drug: methylnaltrexone — Patients will be treated with methylnaltrexone in a standard dosing regimen for their weight: 38-62kg:8 mg, 62-114kg:12 mg, >114 kg: 0.15 mg/kg) Methylnaltrexone will be administered subcutaneously every other day for up to 7 doses.

SUMMARY:
Methylnaltrexone for the treatment of opioid-induced constipation in the setting of palliative or hospice care, is significantly more effective than placebo (1). However, in both the randomized and the open-label phase of the multi center trial showing this favorable outcome, the drug produced rescue-free laxation in only about half of the patients (2). There may be several reasons for this result, since constipation in palliative care patients often has multiple simultaneously occurring causes.

Assuming that constipation of the non-responders is still opioid-induced, one of the possible reasons for not responding to methylnaltrexone could be that central actions of opioids contribute to constipation by reducing motility of the intestines through direct actions in the spinal dorsal horn (2). However, as methylnaltrexone is a µ-receptor antagonist and not all opioids are solely µ-receptor agonists another reason may well be that successful laxation is determined by the receptor-profile of the specific opioid the patient is using.

Opioids do not only influence bowel functioning, but also immune system functioning and angiogenesis. Methylnaltrexone possibly antagonizes these changes, therefore this study will also investigate the influence of methylnaltrexone on immunologic and angiogenic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Receiving palliative care
* Life expectancy ≥ 2 weeks
* Able to give informed consent
* Receiving opioid treatment with either morphine sulphate, oxycodone or fentanyl
* Opioid treatment, both

  * On a regular schedule (not just as needed or rescue doses) for the control of pain or dyspnea for at least 2 weeks before the first dose of methylnaltrexone, and
  * On a stable opioid regimen for at least 3 days before the first dose of methylnaltrexone. This is defined as no dose reduction of ≥ 50%, dose increases are permitted. If rescue medication is prescribed of a different type of opioid than the regular dosed opioid, the rescue medication should be switched to the same type as the regular dosed opioid for at least 3 days before the first dose of methylnaltrexone.
* Has diagnosis of constipation, defined as either

  * < 3 bowel movements during the previous week by history and no clinically notable laxation* in the 24 hours before the first dose of methylnaltrexone, or
  * No clinically notable laxation* in the 48 hours before the first dose of methylnaltrexone.
* Constipation is defined as opioid induced, determined by investigator
* On stable laxative regimen for ≥ 3 days before the first dose of methylnaltrexone. This is defined as at least one type of laxative in an adequate dosing regimen, (e.g. macrogol 2 packets daily, magnesium(hydr)oxide 500 mg three times daily, bisacodyl 10 mg daily or sennoside A+B 10 ml daily) or at least two types of laxatives in a suboptimal dose with patient characteristics hampering optimal treatment.
* If the subject is a woman with presumed child bearing potential; negative urine pregnancy test at screening
* Surgically sterile or agrees to use a medically acceptable method of birth control or practice sexual abstinence for the duration of the methylnaltrexone treatment and the following 15 days. ~

  * including laxation after rescue laxative or enema ~ not necessary for postmenopausal women

Exclusion Criteria:

* Previous treatment with methylnaltrexone
* Known or suspected mechanical gastrointestinal obstruction
* Presence of an other cause of bowel dysfunction that is considered to be a major contribution to the constipation according to investigator
* Presence of a peritoneal catheter for intraperitoneal chemotherapy or dialysis
* Clinically relevant active diverticular disease
* History of bowel surgery within 10 days before first dose of methylnaltrexone
* Fecal ostomy
* Use of vinca alkaloids within previous 4 months
* Body weight <38 kg
* Renal failure defined as EGFR <30 ml/min per 1.73m2 or requires dialysis.
* Known or suspected allergy to methylnaltrexone or similar compounds (e.g. naltrexone or naloxone)
* Participation in a study with investigational products within 30 days before first dose of methylnaltrexone.
* Pregnant or nursing
* Clinically important abnormalities that may interfere with participation or compliance to the study, determined by investigator

Additional exclusion criteria for the immunologic and angiogenic analysis part of the study:

* Chemotherapy or treatment with tyrosine kinase inhibitor during 4 weeks before inclusion or treatment scheduled during participation in this study.
* Treatment with high dose corticosteroids during 2 weeks before inclusion in this study. This is defined as the equivalent of 30 mg of prednisone per day for ≥ 2 consecutive days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving palliative care who are being treated with opioids for symptoms of pain or dyspnea, suffering from constipation, that is not relieved by first line oral laxatives.
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2012-07; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Rescue-free laxation response | Within 4 hours after at least 2 of the first 4 doses (the first week of treatment).
  The proportion of subjects that has a rescue-free laxation response within 4 hours after at least 2 of the first 4 doses (the first week of treatment).

SECONDARY OUTCOMES:
Time to first laxation | Between dosing and day 14
  Time to first laxation after initiation of treatment
Number of laxations | Between dosing and day 14
  * Number of laxations per week
  * Change in BFI score between day 0 and 14
Laxation within 4 hours | Between dosing and day 14
  Presence of laxation within four hours after initiation of treatment
laxation within 4 hours after each dose | Between dosing and day 14
  Number of doses after which laxation occured within four hours after treatment administration
laxation within 24 hours after each dose | Between dosing and day 14
  Number of doses after which laxation occured within 24 hours after treatment administration
laxation within 4 hours after 4 out of 7 doses | Between dosing and day 14
  Did laxation occur within 4 hours after at least 4 out of 7 treatment administrations?

OTHER OUTCOMES:
Changes in leukocyte subsets | Day 0 to day 42
  The concentration of the following markers will be evaluated: T-, B-, NK-cells, monocytes/macrophages, DC subsets, neutrophilic granulocytes, and regulatory cell populations (invariant NKT cells, CD4+CD25+FOXP3+ regulatory T cells.
Changes in serum cytokine levels | Day 0 to day 42
  Changes serum cytokine levels. The concentration of the following markers will be evaluated: IFN-γ, IL-2, IL-4, IL-10, IL-6 and TNF-α.
Determination of the angiogenic profile. | Day 0 to day 42
  * Determination of the angiogenic profile by determination of angiogenic factor blood concentrations and the systemic levels of endothelial progenitor cells.
Determination of the angiogenic potential | Day 0 to day 42
  * Determination of the angiogenic potential of blood on in vitro endothelial cell proliferation assays before and during treatment with methylnaltrexone (in a subgroup of patients, maximally n = 10 per group).

CONTACTS AND LOCATIONS:
Overall Officials: Henk WM Verheul, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (6):
- Netherlands (6):
  - Medical Center Alkmaar, Alkmaar
  - VU University Medical Center, Amsterdam
  - Hospice Demeter, De Bilt
  - Hospice Bardo, Hoofddorp
  - Spaarne Ziekehuis, Hoofddorp
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Derived] Neefjes ECW, van der Wijngaart H, van der Vorst MJDL, Ten Oever D, van der Vliet HJ, Beeker A, Rhodius CA, van den Berg HP, Berkhof J, Verheul HMW. Optimal treatment of opioid induced constipation in daily clinical practice - an observational study. BMC Palliat Care. 2019 Mar 29;18(1):31. doi: 10.1186/s12904-019-0416-7. PMID 30922276
- [Derived] Neefjes EC, van der Vorst MJ, Boddaert MS, Zuurmond WW, van der Vliet HJ, Beeker A, van den Berg HP, van Groeningen CJ, Vrijaldenhoven S, Verheul HM. Clinical evaluation of the efficacy of methylnaltrexone in resolving constipation induced by different opioid subtypes combined with laboratory analysis of immunomodulatory and antiangiogenic effects of methylnaltrexone. BMC Palliat Care. 2014 Aug 20;13:42. doi: 10.1186/1472-684X-13-42. eCollection 2014. PMID 25165428